CLINICAL TRIAL: NCT02467972
Title: Functional Ingredients: Effect in Satiety and Intestinal Health
Brief Title: Functional Ingredients: Effect in Gastrointestinal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Eliana Bistriche Giuntini, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEPFCF194 CEPFCF18; CONEP Brasil (Registry Identifier: CAAE 0042.0.018.000-11); CONEP Brasil (Registry Identifier: CAAE 0069.0.018.198-11)
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Overweight; Diabetes; Constipation
Keywords: Hunger and satiety; Hormones gastrointestinal; Bowel movements
MeSH Terms: conditions — Overweight; Diabetes Mellitus; Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- UBF group (Experimental): Ready-to-eat frozen soups added unripe banana flour (18 portions; 3 times/week)
  Interventions: Dietary Supplement: Ready-to-eat frozen soups added unripe banana flour
- Control (Placebo Comparator): Ready-to-eat frozen soups added maltodextrin (18 portions; 3 times/week)
  Interventions: Dietary Supplement: Ready-to-eat frozen soups added maltodextrin
- Inulin group (Experimental): Ready-to-eat frozen soups added inulin (18 portions; 3 times/week)
  Interventions: Dietary Supplement: Ready-to-eat frozen soups added inulin
- Nisin group (Experimental): Ready-to-eat frozen soups added nisin (18 portions; 3 times/week)
  Interventions: Dietary Supplement: Ready-to-eat frozen soups added nisin

INTERVENTIONS:
Dietary Supplement: Ready-to-eat frozen soups added unripe banana flour — Ready-to-eat frozen soups added unripe banana flour (18 portions; 3 times/week)
  Arms: UBF group
Dietary Supplement: Ready-to-eat frozen soups added maltodextrin — Ready-to-eat frozen soups added maltodextrin (18 portions; 3 times/week)
  Arms: Control
Dietary Supplement: Ready-to-eat frozen soups added inulin — Ready-to-eat frozen soups added inulin (18 portions; 3 times/week)
  Arms: Inulin group
Dietary Supplement: Ready-to-eat frozen soups added nisin — Ready-to-eat frozen soups added nisin (18 portions; 3 times/week)
  Arms: Nisin group

SUMMARY:
The addition of fructans or unripe banana flour to frozen meals can change the hormonal parameters related to hunger and satiety, improve the bowel movements and increase in colonic bacteria population measured by microbiological determinations (qPCR). The inulin no can change bowel movements and increase in colonic bacteria population measured by microbiological determinations (qPCR)

DETAILED DESCRIPTION:
Non-transmissible chronic diseases have been constantly related to the consumption of diets with inadequate nutrient input; at the same time, the ingestion of unavailable carbohydrates have presented an inverse relationship with the risk for these diseases. Among these carbohydrates is inulin, a fructan considered as a prebiotic and the unripe banana flour, rich in resistant starch, which may contribute to the intestinal health.

This study evaluated the effect of regular intake of frozen soups added functional ingredients (fructans and unripe banana flour) by heath volunteers, about gastrointestinal hormones, satiety and bowel movements.

ELIGIBILITY:
Inclusion Criteria:

- good health condition

Exclusion Criteria:

* history of renal or gastrointestinal disease
* hyperthyroidism
* diabetes, nor parents with diabetes
* for women: not pregnant, breastfeeding or using hormonal therapy
* using any drug that might affect the digestion of food and absorption (antibiotics, laxatives)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in hormonal parameters related to hunger and satiety. | 6 weeks
  Changes in satiety measured by specific hormones kit
Change in bowel function | 6 weeks
  Changes measured by GSRS and daily questionnaires
Change in colonic bacteria population | 6 weeks
  Changes measured by microbiological analysis by r16SDNA sequencing
Change in satiety | 6 weeks
  Changes in satiety measured by Visual Analogue Scale questionnaire.

SECONDARY OUTCOMES:
Change in biochemical parameters | 6 weeks
  Changes measured by biochemical kit

CONTACTS AND LOCATIONS:
Overall Officials: Elizabete W Menezes, Prof Assoc, Principal Investigator — Faculty of Pharmaceutical Sciences of University of Sao Paulo
Locations (1):
- Faculty of Pharmaceutical Sciences USP, São Paulo, São Paulo, Brazil